CLINICAL TRIAL: NCT02244385
Title: Manchester Antenatal Vascular Service
Acronym: MAViS
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11/NW/0426
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Vascular Disease
Keywords: vascular disease; pregnancy; chronic hypertension; diabetes; obesity
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood sample Urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: No intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
25-30% of women with preexisting vascular disease (chronic hypertension/diabetes/obesity) will develop pre-eclampsia and or growth restriction. In addition, the frequency of stillbirths in this group is dramatically increased over the general population. Pregnancy complications in this very heterogeneous group are likely to be a combination of a failure of the maternal vasculature to adapt to pregnancy and/or a failure of placental development. The relative contribution of these two mechanisms is poorly understood and current preventative strategies (aspirin) in this group only prevent a small number of adverse outcomes. This important and complex group have been inadequately investigated to date mainly because of the diversity of their underlying disease complicating prospective research studies.

The evolution of tools which allow more detailed assessments of both uteroplacental blood flow and maternal vascular function will enable us to perform prospective studies in these women and to develop targeted preventative measures. Recent biomarker studies have also identified a number of biomarkers which have not yet been assessed in these high risk groups.

ELIGIBILITY:
Inclusion Criteria:

Women with preexisting vascular disease:

1. chronic hypertension BP ≥140/90 at ≤14 weeks
2. chronic hypertension requiring antihypertensive treatment ≤ 14 weeks
3. pre gestational diabetes with evidence of vascular complications (hypertension, nephropathy)
4. history of ischemic heart disease
5. previous early onset pre-eclampsia (delivery < 32 weeks)
6. Obesity (BMI ≥ 40) with any history of hypertension or booking BP≥130/80

Exclusion Criteria:

Women who do not meet the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women will be approached about the study in a dedicated clinic run within the Maternal & Fetal Health Research Centre.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2011-07; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | At recruitment (<14 weeks gestation) and at 16-18 weeks, 22-26 weeks & 30-34 weeks gestation

SECONDARY OUTCOMES:
Vascular compliance | At recruitment (<14 weeks gestation) and at 16-18 weeks, 22-26 weeks & 30-34 weeks gestation
Uteroplacental assessment | At recruitment (<14 weeks gestation) and at 16-18 weeks, 22-26 weeks & 30-34 weeks gestation

OTHER OUTCOMES:
urinary albumin | At recruitment (<14 weeks gestation) and at 16-18 weeks, 22-26 weeks & 30-34 weeks gestation
Urinary podocyte markers | At recruitment (<14 weeks gestation) and at 16-18 weeks, 22-26 weeks & 30-34 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Myers, PhD MRCOG BM BS, Principal Investigator — University of Manchester
Locations (1):
- Maternal & Fetal Health Research Centre, 5th Floor St Mary's Hospital, Manchester, United Kingdom